CLINICAL TRIAL: NCT02449694
Title: Single-arm Prospective Trial to Evaluate The Safety and Performance of The Portable Organ Care System (OCS™) Liver For Preserving and Assessing Donor Livers for Transplantation
Brief Title: Trial of the TransMedics Organ Care System™ Liver For Preserving and Assessing Donor Livers for Transplantation
Acronym: REVIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-LVR-022015
Record Dates: First submitted 2015-05-11; First posted 2015-05-20 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Liver Preservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OCS Liver (Experimental): OCS Liver will be used to preserve the donor liver
  Interventions: Device: OCS Liver

INTERVENTIONS:
Device: OCS Liver — OCS Liver will be used to preserve the donor liver

SUMMARY:
A prospective, single-center controlled trial to evaluate the safety and performance of the portable Organ Care System (OCS) Liver for preservation and assessment of donor livers for transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Registered male or female primary Liver transplant candidate
* Age ≥18 years old
* Signed: written informed consent

Exclusion Criteria:

* Acute, fulminant liver failure;
* Prior solid organ or bone marrow transplant;
* Chronic use of hemodialysis or diagnosis of chronic renal failure, defined as chronic serum creatinine of >3 mg/dl (>265 mmol/L) for >2 weeks and/or requiring hemodialysis;
* Multi-organ transplant;
* Ventilator dependent;
* Dependent on > 1 IV inotrope to maintain hemodynamics;
* Malignancy excluding HCC;
* Infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05; Primary Completion 2017-09-19 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of donor livers preserved by OCS in a near physiologic state. | Within 1 day of organ retrieval
Number of events directly related to the use of the OCS Liver that led to the donor liver being deemed not clinically acceptable and, as a result, not transplanted | Within 1 day of organ retrieval

SECONDARY OUTCOMES:
Number of donor livers maintained in a metabolically active and functioning state during preservation. | Within 1 day of organ retrieval
Number of donor livers monitored for perfusate temperatures, SvO2, hematocrit, Hepatic Artery flow rates, Portal Vein flow rate, Hepatic Artery pressure, Portal vein pressure, and bile production during preservation. | Within 1 day of organ retrieval
Frequency of liver graft-related serious adverse events | 30 days after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- St. James's University Hospital, Leeds, West Yorkshire, United Kingdom